CLINICAL TRIAL: NCT04533698
Title: Impact of Fluid Resuscitation Protocol on the Incidence of Reoperation for Bleeding After Emergency Cardiopulmonary Bypass Grafting
Acronym: Volu-CABG
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Principal Investigator, Alexa Hollinger, Principal Investigator, University Hospital, Basel, Switzerland
Other Study IDs: 2020-01833
Record Dates: First submitted 2020-08-26; First posted 2020-08-31 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Resternotomy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Resternotomy
  Interventions: Other: Assessment of reason for resternotomy
- No resternotomy
  Interventions: Other: Assessment of reason for avoidance of resternotomy

INTERVENTIONS:
Other: Assessment of reason for resternotomy — No intervention is performed. Reasons for resternotomy (coagulation, fluid balance and other) are retrospectively assessed.
  Groups: Resternotomy
Other: Assessment of reason for avoidance of resternotomy — No intervention is performed. Reasons for avoidance resternotomy (coagulation, fluid balance and other) are retrospectively assessed.
  Groups: No resternotomy

SUMMARY:
This is a retrospective data analysis of patients that underwent elective or emergency cardiopulmonary bypass. Resternotomy due to bleeding is frequent after sternotomy. Also due to implementation of Argipressin into clinical practice fluid resuscitation protocol has changed to more vasopressors and less fluid within the past five years. The investigators want to explore the influence of volume resuscitation protocol on incidence of rethoracotomy during the past twenty years.

ELIGIBILITY:
Inclusion Criteria:

* All patients that underwent elective or emergency aortocoronary bypass at the University Hospital Basel between 2009 and 2020.

Exclusion Criteria:

* None.

Ages: 18 Years to 99 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients that underwent elective or emergency aortocoronary bypass.
Sampling Method: Non-Probability Sample
Enrollment: 265 (Actual)
Dates: Start 2009-01-01 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Resternotomy | 7 days
  Resternotomy yes or no after elective or emergency aortocoronary bypass

REFERENCES:
- [Derived] Bruno J, Varayath M, Gahl B, Miazza J, Gebhard CE, Reuthebuch OT, Eckstein FS, Siegemund M, Hollinger A, Santer D. Conservative fluid resuscitation protocol does not reduce the incidence of reoperation for bleeding after emergency CABG. Sci Rep. 2024 Sep 9;14(1):21037. doi: 10.1038/s41598-024-71028-8. PMID 39251616